CLINICAL TRIAL: NCT02375126
Title: Normal Quantitative EEG (qEEG) Dataset for the Use in Comparison With Patients Suffering Carbon Monoxide (CO) Poisoning
Brief Title: Normal Quantitative EEG (qEEG) Dataset
Acronym: NormalEEG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 1024985
Record Dates: First submitted 2015-02-19; First posted 2015-03-02 (Estimated); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Carbon Monoxide Poisoning
MeSH Terms: conditions — Carbon Monoxide Poisoning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Ages 18-35, no antidepressant use: Ages 18-35, up to 15 males and 15 females, no antidepressant use
  Interventions: Procedure: Electroencephalography
- Ages 36-55, no antidepressant use: Ages 36-55, up to 15 males and 15 females, no antidepressant use
  Interventions: Procedure: Electroencephalography
- Ages 18-55, with antidepressant use: Ages 18-55, up to 10 males and 10 females, taking antidepressants
  Interventions: Procedure: Electroencephalography

INTERVENTIONS:
Procedure: Electroencephalography — Electroencephalography (EEG) is a relatively inexpensive measurement of basic brain activity. Traditional EEG techniques rely on the clinician to visually examine the electrical current waveforms to identify abnormal signal patterns and slowing. Abnormalities on EEG have been reported following CO poisoning, though the literature is scarce. While current EEG technologies record EEG signals digitally, rather than writing directly to paper, computer-assisted analysis of the data (quantitative EEG, or qEEG) has not been widely embraced, in part because clinicians are unsure what patterns revealed by computer-assisted analysis represent abnormal activity.
  Other Names: EEG

SUMMARY:
In this study, the investigators will collect EEG data in normal, healthy volunteers without a history of prior brain injury. This data will be analyzed by computer (quantitative, or qEEG) and stored in a normative database so that, in the future, the investigators can better understand and characterize the brain damage that can result from carbon monoxide (CO) poisoning and other types of brain injury.

DETAILED DESCRIPTION:
This is a pilot, prospective, non-comparative, non-invasive, minimal risk research study to obtain qEEG data on normal, healthy individuals to include in a normal control database for use in comparison with patients with CO poisoning and other types of brain injury. The use of anti-depressant medication use is relatively common in the general adult population. There is varying opinion whether anti-depressant medication alters an otherwise normal clinical EEG. We have included healthy individuals taking anti-depressant medication to determine if those medications influence the EEG. The EEG data will be collected, analyzed, and stored for use in future research studies and for clinical care. Evaluating patients with qEEG methodology may assist in diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, from 18 to 55 years old at the time of study enrollment. Women who are greater than 6 weeks post-partum, who are breastfeeding are allowed to participate if they are able to finish the electroencephalography (EEG) without interruption.
* Able to speak and read English as their primary language.
* Agrees to, and appears able to, participate in all outcome assessments.
* Demonstrates the ability to offer informed consent and signs the study informed consent document.

Exclusion Criteria:

* Vulnerable populations including, prisoners, pregnant women, and minors.
* Women who are less than 6 weeks post-partum.
* Unwilling or unable to participate in planned study visits.
* Any past history of brain injury due to trauma, surgery, hypoxia, infection, inflammation, toxicity (e. g., carbon monoxide poisoning), or cerebrovascular etiology.
* Individuals with a diagnosis of, or a persistent history of, or symptoms of a neurological disorder (e.g., tinnitus, vertigo, chronic fatigue, numbness, tingling, chronic migraine, fibromyalgia, multiple sclerosis).
* Currently undergoing therapy for affective disorders, behavioral disorders, or psychological disorders.
* Diagnosis of post-traumatic stress disorder or sub-clinical post-traumatic stress symptoms.
* Diagnosis of diabetes mellitus, type 1 and type 2.
* Current complaints of brain injury symptoms such as cognitive or affective problems.
* Known neuroimaging abnormalities.
* Participants taking daily prescription drugs or oral over the counter medications beyond vitamins that could impact a normal outcome determined by the Principal Investigator (e.g., beta blockers).
* Participants who are ≥45 may be taking statins or angiotensin converting enzyme (ACE) inhibitors.
* Participants between the ages of 18-55 may be taking antidepressants indicated for depression or post-partum depression.
* Oral or injectable contraceptives are permitted
* Known atrial septal defect, including but not limited to patent foramen ovale.
* History of bypass surgery.
* History of hydrocephalus/microcephaly/macrocephaly.
* History of developmental delay or learning disorder as a child.
* Previous or current use of any illicit drug, at any age.
* Current positive urine drug test for any illicit substance.
* History, by self-report in the last year, of alcohol abuse.
* Current or previous tobacco use, with the exception of minimal use during adolescence.
* Use of any assistive hearing device, or unable to verbally communicate due to hearing loss.
* History, by self-report, of receiving chemotherapy drugs or therapeutic ionizing radiation to the head.
* Foreign material in the head.
* Active malignancy or prior malignancy (except basal cell carcinoma) within the last 5 years.
* Unable to abstain from caffeine products for at least a 2 hour interval.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Normal, healthy volunteers (adult men and women, ages 18-55) will be selected from a carefully screened convenience sample.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Electroencephalography Completion Questionnaire (Y/N) | Baseline
  Electroencephalography study completed for the participant. (Y/N)

CONTACTS AND LOCATIONS:
Overall Officials: Lindell K Weaver, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Healthcare, LDS Hospital, Salt Lake City, Utah, United States